CLINICAL TRIAL: NCT06516614
Title: Sleep Promoting Intervention to Improve Diabetes Outcomes and Executive Function in Adolescents With T1D
Brief Title: Sleep Coach for Adolescents With Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Sarah Jaser, Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 230074
Record Dates: First submitted 2024-07-17; First posted 2024-07-24 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep-Promoting Intervention (Experimental): Individualized sleep-promoting program for adolescents with type 1 diabetes
  Interventions: Behavioral: Sleep Coach
- Enhanced Usual Care (Active Comparator): Educational Materials
  Interventions: Behavioral: Diabetes Education

INTERVENTIONS:
Behavioral: Sleep Coach — Sleep-promoting intervention consisting of 4 phone sessions to improve sleep duration and consistency.
  Arms: Sleep-Promoting Intervention
Behavioral: Diabetes Education — Participants will receive a a binder with educational information about diabetes and educational messages from the study team.
  Arms: Enhanced Usual Care

SUMMARY:
The goal of this work is to conduct a randomized trial evaluating the effects of a behavioral intervention to increase sleep duration and quality for adolescents with type 1 diabetes (T1D). The impact of the sleep-promoting intervention on executive function and glycemic outcomes will be assessed. We will also explore multiple components of the recently identified central nervous system glymphatic system and evaluate how these components change and impact brain integrity and function with improved sleep.

DETAILED DESCRIPTION:
This randomized controlled trial will assess whether a behavioral coaching intervention to improve sleep duration and quality in adolescents with type 1 diabetes will improve glucose control and executive function. We will recruit a sample of 150 adolescents with type 1 diabetes (T1D) and their caregivers at a single medical center. We plan to recruit equal numbers of boys and girls and over-enroll youth from minoritized racial and ethnic groups. After obtaining informed consent/assent and baseline data, we will randomize adolescents to the Sleep Coach condition (n=75) or the Enhanced Usual Care condition (n=75). Randomization will be computerized, and adolescents will be stratified by diabetes device use (insulin pumps, continuous glucose monitors) and age (11-14 years vs. 15-17 years). Adolescents and caregivers will complete survey measures again at 3 months, 6 months, and 12 months during regularly scheduled clinic visits. Adolescents will complete the NIH Toolbox measures of executive function at each study visit. Adolescents will be asked to wear a FitBit watch to assess sleep and complete sleep diaries at baseline and 3 months.

Participants randomized to the Sleep Coach group will be sent a binder with intervention materials for the 4 sessions. They will schedule individual phone calls with a trained member of the research team at a convenient time. The first call is expected to last 20-30 minutes, and the other calls are expected to last 10-15 minutes. Caregivers will receive an overview of the sleep intervention content, and they will be asked to support adolescents' attempts to change sleep habits.

Adolescents randomized to Enhanced Usual Care will receive diabetes education materials developed by our team for adolescents with T1D (based on publicly available materials on diabetes.org). Printed materials will be sent via mail and content will be shared via smart phone messages on the same schedule as participants randomized to the Sleep Coach intervention.

A representative group of 50 of the 150 adolescents in the study will be invited to participate in an additional study visit prior to the intervention to obtain magnetic resonance imaging (MRI) of the brain. Adolescents who agree to complete MRI of the brain will be asked to complete a follow-up visit approximately 6 months after the baseline visit, following the same protocol, and they will complete the daily sleep diary questions and share sleep data for another week.

ELIGIBILITY:
Inclusion Criteria:

* 11-17 years of age at the time of enrollment
* Diagnosed with type 1 diabetes for ≥ 12 months
* Report insufficient sleep (< 8 hrs./night for 13-17 year-olds, <9 hrs./night for 11-12 year-olds) but have no other sleep disorders or sleep apnea
* Are not meeting the target for HbA1c (<7%)
* Able to read /speak English

Exclusion Criteria:

* Participant has other serious health conditions that interfere with diabetes management
* Optional MRI portion of the study - anything that would prevent an adolescent from receiving a high-quality MRI of the brain (metal implants or inability to hold still for an MRI which may take up to 60 minutes)

Inclusion criteria for caregivers:

* Currently living with the child (at least 50% of the time)
* Speak and read English

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Sleep Duration | 3 months
  Total Sleep Time (average minutes per night) measured with Fitbit over 7 nights
Sleep Variability | 3 months
  Individual difference in sleep duration (minutes) measured with Fitbit over 7 nights

SECONDARY OUTCOMES:
Executive Function BRIEF2 | 12 months
  Behavior Rating Inventory of Executive Function 2nd Edition: 63-item measure, completed by parents to assess adolescent executive function in their daily life. Higher Global Executive Composite score indicates better executive function.
NIH Toolbox Dimensional Card Sort Test | 12 months
  Dimensional Change Card Sort Test takes 4 minutes for adolescents to complete on an iPad, assesses inhibition, a component of executive function
NIH Toolbox List Sorting Working Memory Test | 12 months
  List Sorting Working Memory takes 8-10 minutes for adolescents to complete on an iPad, assesses working memory, a component of executive function
Diabetes Management - Adolescent Report | 12 months
  Self-Care Inventory-Short Form: 9-item measure, assesses key components of adolescent diabetes management. Higher mean scores indicate better diabetes self-care.
Diabetes Management - Parent Report | 12 months
  Self-Care Inventory-Short Form: 9-item measure, assesses key components of adolescent diabetes management. Higher mean scores indicate better diabetes self-care.
Sleep Quality | 12 months
  Pittsburgh Sleep Quality Index (PSQI): 21-item measure completed by adolescents, assesses sleep quality. Higher scores indicate poorer sleep quality.
Hemoglobin A1C | 12 months
  An indicator of average blood glucose levels. HbA1c is collected as part of usual care and will be extracted from adolescents' medical records
Time in Range | 12 months
  Blood glucose levels, measured with continuous glucose monitors, that are within the target range (70-180 mg/dL) over 14 days. Time in Range is reported as a percentage and higher levels indicate better glycemic control.
Magnetic Resonance Imaging (MRI) of Brain: Glymphatic Flow | 6 months
  Fluid motion along perivascular spaces is assessed from MRI of the brian
Fractional Anisotropy from MRI of the Brain | 6 months
  Fractional anisotropy is calculated from diffusion tensor imaging MRI. Higher FA is associated with better white matter integrity in the brain

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Jaser, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States